CLINICAL TRIAL: NCT03234361
Title: Preventing Hypertension and Sympathetic Overactivation by Targeting Phosphate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU 012017-052
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Hypertension
Keywords: Hypertension; High phosphorus diet; FGF 23; 24 hour ambulatory blood pressure; Muscle sympathetic nerve
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Phosphate Phase (Experimental): All subjects will be on a low Pi diet containing 700mg/day of phosphate and 2 capsules of sodium phosphate with 500mg/day of phosphate for 4 weeks.
  Interventions: Dietary Supplement: High Phosphate Phase
- Low Phosphate Phase (Placebo Comparator): All subjects will be on a low Pi diet containing 700mg/day of phosphate and 2 capsules of sodium chloride for 4 weeks.
  Interventions: Dietary Supplement: Low Phosphate Phase

INTERVENTIONS:
Dietary Supplement: High Phosphate Phase — 2 capsules of sodium phosphate with 500mg/day of phosphate.
  Arms: High Phosphate Phase
Dietary Supplement: Low Phosphate Phase — 2 capsules of sodium chloride.
  Arms: Low Phosphate Phase

SUMMARY:
An increasing number of studies have indicated that most fast food and common grocery items, contain large amount of inorganic phosphate-based food additives , which are highly absorbable. The long-term cardiovascular consequences of a high phosphate diet are unknown but the existing database implicates phosphate excess as an independent risk factor for cardiovascular events in individuals with and without chronic kidney diseases (CKD). High phosphate consumption clearly induces BP elevation in rats with normal kidneys. However, the mechanisms underlying phosphate-induced hypertension and the relevance of these rodent studies to human hypertension have not been determined. We seek to investigate the role of high phosphate diet in human hypertension and assess the effect of high phosphate diet on muscle sympathetic nerve activity and the exercise pressor reflex.

DETAILED DESCRIPTION:
Animal studies suggest that high phosphate diet raises blood pressure but the mechanism underlying this phenomenon is not known. To study the effect of high phosphorus diet on blood pressure in humans, we will perform randomized crossover studies in stage 1 prehypertensive subjects. To ensure stable Pi intake prior to randomization, Pi consumption will be estimated by food recall during a run-in and washout phase for 2 consecutive days, using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool (https://epi.grants.cancer.gov/asa24/). After the run-in period, all subjects will be maintained on a low Pi diet (700 mg/d) and a low Na diet of approximately 1,930 mg/d throughout the study for 8 weeks. Subjects will also be randomized to receive Sodium Phosphate 2 capsules daily (containing a total of 500 mg of Pi, 372mg of sodium) for 4 weeks during the high Pi phase (total Pi intake 1,200 mg/d) vs 2 capsules of Sodium Chloride (NaCl, containing a total of 372mg of sodium) to match Na content to Sodium Phosphate without extra Pi daily for 4 weeks during the low Pi phase (total Pi intake = 700 mg/d).

The total Na intake during the entire study will be at recommended level of 2,300 mg/d. Investigational drug service at UT Southwestern will dispense Sodium Phosphate vs. NaCl tablets tablets and the study subjects will be blinded to the type of supplement they receive.

During the periods of high and low Pi phases, we will monitor 24-hr UPiV to ensure adherence. Since approximately 70% of ingested Pi is absorbed and excreted in the urine, we expect 24-hr UPiV excretion to be approximately 840 mg during the high Pi phase and 490 mg during the low Pi phase. If 24-hr UPiV is < 800 mg during the high Pi diet or > 500 mg during the low Pi diet, the research dietitian will provide additional counseling to improve adherence to the menu plan. If needed, the research diet will be altered to be more compatible with subject preference. 24-hr UPiV will be reassessed within 1 week in these individuals. If the levels remain below goal, subjects will be excluded from the study.

24-hr urinary Pi, Na, K, Cr, and Ca excretion will be assessed after weeks 2 and 4 of the low and high Pi phases. Serum electrolytes and Pi will be monitored every 2 weeks. Serum FGF23, PTH, and soluble Klotho levels and 24-h ambulatory BP will be obtained after 4 weeks on the study diet. Then, on a separate day, we will assess muscle SNA and BP at rest and during rhythmic handgrip of 30% and 45% each for 3 minutes. Additionally, we will test the role of dietary Pi on the response to isometric exercise by assessing SNA and BP during static handgrip at 30% MVC for 2 minutes followed by post exercise circulatory arrest (PECA). The latter maneuver will maximally activate the metaboreflex. Each exercise intervention will be separated by at least 30 minutes. The order of exercise intervention will be randomized. Subsequently, subjects will stop the first study supplement and undergo washout for 2 weeks. After 2 weeks of washout, they will receive the 2nd study supplement. Measurement of 24-h ambulatory BP, SNA at rest and during handgrip exercise will be repeated in the same fashion.

ELIGIBILITY:
Inclusion Criteria: (answer must be yes to all to enter trial; check yes or no)

º ≥ 18 years of age

º Stage 1 Prehypertension (office BP 120-129/80-84 mmHg and normal ABPM <130/80)

Exclusion Criteria: (answer must be no to all to enter trial)

º Diabetes mellitus or other systemic disease

º Cardiopulmonary disease

º Treatment with antihypertensive medications

º eGFR< 60 ml/min/1.73m2

º Pregnancy

º Hypersensitivity to nitroprusside or phenylephrine

º Psychiatric illness

º H/o substance abuse or current smoker

º H/o malignancy

º Serum Phos <2.4 mg/dL or >4.5 mg/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
24-hour Blood Pressure measured by Ambulatory Blood Pressure Monitor. | 4 weeks
  Blood pressure will be measured through an ambulatory blood pressure monitoring device by Space Labs # 90217, worn by each participant after completing each phase, This will suggest if participant's blood pressure increased during high phosphorus phase as compared to low phosphorus phase.

SECONDARY OUTCOMES:
Muscle Sympathetic Nerve Activity (MSNA) | 4 weeks after high phosphorus and 4 weeks after low phosphorus diet
  MSNA will be measured during both diet phases using microelectrodes inserted in the peroneal nerve. This will assess the impact of phosphate intake on MSNA.

CONTACTS AND LOCATIONS:
Overall Officials: Wapen Vongpatanasin, MD, Principal Investigator — UT southwestern
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sullivan CM, Leon JB, Sehgal AR. Phosphorus-containing food additives and the accuracy of nutrient databases: implications for renal patients. J Ren Nutr. 2007 Sep;17(5):350-4. doi: 10.1053/j.jrn.2007.05.008. PMID 17720105
- [Background] Benini O, D'Alessandro C, Gianfaldoni D, Cupisti A. Extra-phosphate load from food additives in commonly eaten foods: a real and insidious danger for renal patients. J Ren Nutr. 2011 Jul;21(4):303-8. doi: 10.1053/j.jrn.2010.06.021. Epub 2010 Nov 5. PMID 21055967
- [Background] Ketteler M, Wolf M, Hahn K, Ritz E. Phosphate: a novel cardiovascular risk factor. Eur Heart J. 2013 Apr;34(15):1099-101. doi: 10.1093/eurheartj/ehs247. Epub 2012 Oct 7. No abstract available. PMID 23045267
- [Background] Karp H, Ekholm P, Kemi V, Itkonen S, Hirvonen T, Narkki S, Lamberg-Allardt C. Differences among total and in vitro digestible phosphorus content of plant foods and beverages. J Ren Nutr. 2012 Jul;22(4):416-22. doi: 10.1053/j.jrn.2011.04.004. Epub 2011 Jul 13. PMID 21741857
- [Background] Suzuki Y, Mitsushima S, Kato A, Yamaguchi T, Ichihara S. High-phosphorus/zinc-free diet aggravates hypertension and cardiac dysfunction in a rat model of the metabolic syndrome. Cardiovasc Pathol. 2014 Jan-Feb;23(1):43-9. doi: 10.1016/j.carpath.2013.06.004. Epub 2013 Aug 8. PMID 23932324
- [Background] Scanni R, vonRotz M, Jehle S, Hulter HN, Krapf R. The human response to acute enteral and parenteral phosphate loads. J Am Soc Nephrol. 2014 Dec;25(12):2730-9. doi: 10.1681/ASN.2013101076. Epub 2014 May 22. PMID 24854273
- [Background] Hu MC, Shi M, Cho HJ, Adams-Huet B, Paek J, Hill K, Shelton J, Amaral AP, Faul C, Taniguchi M, Wolf M, Brand M, Takahashi M, Kuro-O M, Hill JA, Moe OW. Klotho and phosphate are modulators of pathologic uremic cardiac remodeling. J Am Soc Nephrol. 2015 Jun;26(6):1290-302. doi: 10.1681/ASN.2014050465. Epub 2014 Oct 17. PMID 25326585